CLINICAL TRIAL: NCT01388296
Title: Minimum Alveolar Concentrations of Sevoflurane for Maintaining Bispectral Index Below 50 in Morbidly Obese Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Procare Riaya Hospital (Other)
Responsible Party: Principal Investigator, Ahed ZEIDAN, MD, Procare Riaya Hospital
Other Study IDs: PRH 03
Record Dates: First submitted 2011-06-30; First posted 2011-07-06 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Bisbectral index (BIS)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Morbidly obese patients: BMI 40-50 k/m2
- Morbidly obese: BMI 50-60 k/m2
- Morbidly obeses: BMI 60-70 k/m2

SUMMARY:
the target of this study is to assess the minimum alveolar concentration of sevoflurane to maintain theBispectral Index below 50.The minimum alveolar concentration (MAC) for maintaining Bispectral Index below 50 (MACBIS50) of sevoflurane has been reported previously in adult with Body Mass Index ( BMI) < 40 to be 0.97 and in enfant to be 2.83%, However, there is no study assessed theBispectral Index below 50 (MACBIS50 ) in morbidly obese patient (BMI > 40). The first aim of our study is to assess the MACBIS50 of sevoflurane in morbidly obese patients BMI 40 - 70 using the Continuous Reassessment Method (CRM) in 80 % of patients.

DETAILED DESCRIPTION:
After ethical committee approval and written informed consent, 30 morbidly obese adult patients , BMI 40- 70Kg/m², ASA physical status 1 and 2 , aged 18-49 yr, , undergoing elective bariatric surgery under general anesthesia using sevoflurane, were included in this study.

Monitoring consisted of noninvasive blood pressure, Electrocardiogram (ECG) , pulse oximetry, and BIS. All subjects received a standard dose of 2 mcg/kg fentanyl approximately 20 min before induction of general anesthesia. a standard BIS® monitor strip was applied before fentanyl administration and induction of general anesthesia. Induction was performed in all patients with 2m/kg propofol, 0.2 mg/kg cisatracuruim, followed by direct laryngoscopy and tracheal intubation. Therefore, when BIS reached > 65 , sevoflurane was started immediately at the predetermined dose.

The endtidal sevoflurane concentration was adjusted with starting dose for the first cohort patients 1% and maintained for 10 min to ensure equilibration with the cerebral anesthetic partial pressure followed by a 1-min assessment of BIS taken at 10-s intervals. Briefly, a first dose is given to the first patient and the next doses are given according to the following rule: if the subject responds positively (BIS<50), the dose is decreased one step for the next subject, and conversely, if the subject does not respond (BIS>50), the dose is increased one step. The dose adjustment is 0.2% for sevoflurane. The CRM is used to calculate the dose adjustment for every cohort with the number of patients for every cohort .

ELIGIBILITY:
Inclusion Criteria:

* morbidly obese patient
* BMI 40-70
* age : 20-40 year

Exclusion Criteria:

* Age< 20 and > 40
* BMI < 40 and > 70
* comorbidity

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Morbidly obese patients weighting BMI 40-70 k/m2
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Minimal alveolar concentration of Sevoflurane for Maintaining BIS Below 50 | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ahed ZEIDAN, MD, Study Chair — Procare Riaya Hospital
Locations (1):
- Procare Riaya Hospital, Khobar, Estern, Saudi Arabia